CLINICAL TRIAL: NCT02833025
Title: Point-of-care Assessment of Thrombin Generation and Platelet Function in Children Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Point-of-care Assessment of Thrombin Generation and Platelet Function in Children Requiring Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Synapse B.V. Research Institute, University of Maastricht (Unknown)
Responsible Party: Principal Investigator, James O'Leary, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000053849
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Platelet Function Tests; Thrombin Generation Tests; Perioperative Coagulopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thrombin generation and Platelet Function Testing — Point-of-care testing of thrombin generation, platelet function, and rotational thromboelastometry

SUMMARY:
Coagulopathy after cardiopulmonary bypass (CPB) is associated with increased morbidity and mortality. Clot formation and clot stability are important factors in coagulation and hemostasis. As such platelet dysfunction and impaired thrombin generation play a central role in bleeding after cardiac surgery. The primary objective of this study is to evaluate the relationship between point-of-care determined platelet function and thrombin generation and postoperative bleeding in infants and young children undergoing cardiac surgery with cardiopulmonary bypass adjusting for clinically important confounding factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤5 years
2. Undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

1. Non-english speaking parents/care-givers
2. Refusal to consent
3. Extracorporeal membrane oxygenation (ECMO) or ventricular assist device prior to surgery
4. Therapeutic heparin use (unfractionated or low molecular weight) in the immediate preoperative period (<12 hr)
5. Weight <3 kg

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged ≤5 years undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative chest tube blood loss | 24hr

SECONDARY OUTCOMES:
Postoperative chest tube blood loss | 6hr
Postoperative chest tube blood loss | 12hr
Transfusion of blood products | 24hr
All-cause mortality | within 30 days
Length of hospital stay | through study completion, an average of less than one month
Length of ICU stay | within 30 days
Duration of mechanical ventilation | within 30 days
Inotropes | within 30 days
  Duration of inotropic support
Kidney injury | within 30 days
  Acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: James D O'Leary, MBBCh, MM, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No